CLINICAL TRIAL: NCT07135700
Title: Hemodynamic Evaluation and Assessment of DIRECT myocaRdial and Sublingual Capillary Perfusion in Thoracic Surgery Patients on Cardiopulmonary Bypass
Acronym: DIRECT-HEART
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Ufuk Baldan, Resident Cardiac Surgery. MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: DIRECT-HEART
Record Dates: First submitted 2025-08-13; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Microcirculatory Perfusion
Keywords: cardiac surgery; microcirculation; capillary perfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery patients: In order to be eligible to participate in this study, a participant must meet all of the following criteria:
  * Adult patients (18 years or older)
  * Use of central cannulated CPB through median sternotomy
  * Patients undergoing valve surgery or a supracoronary ascending aorta replacement
  * Good LVEF and RVF
  * LAVI < 50 ml/m2, and right atrial volume index (RAVI) < 45 ml/m2,

SUMMARY:
After cardiac surgery, some people may experience problems with their circulation or how well the heart pumps. This can occur because the smallest blood vessels in the heart do not function properly. When these vessels don't work correctly, organs and tissues don't receive enough oxygen and nutrients, which can lead to circulatory problems and organ damage.

Typically, treatments focus on improving the larger blood vessels, such as blood pressure and heart function, but the investigators don't yet know enough about the smallest blood vessels. In this study, the investigators measure blood flow using a special camera (a microscope) at two locations: under the tongue and directly on the heart. Measurements under the tongue are already performed more frequently, but measurements directly on the heart are still new.

If the investigators can demonstrate that differences in cardiac blood flow can also be observed under the tongue, it will become easier to conduct research on microcirculation. The use of the device is safe, and measurements are performed under strict supervision and control by experienced physicians and researchers.

Ultimately, the investigators hope to use this knowledge to better prevent or treat complications after cardiac surgery.

The aim of this research is to investigate whether measurements of blood flow in the smallest blood vessels (microcirculation) on the heart provide the same information as measurements of microcirculation under the tongue.

This appears to be describing a clinical study comparing sublingual and epicardial microcirculation monitoring techniques to potentially establish a less invasive method for assessing cardiac microvascular function in post-surgical patients.

DETAILED DESCRIPTION:
Congruence of micro- and macrocirculation is essential in participants during the postcardiotomy period to maintain hemodynamic stability [1,2]. At the capillary (i.e. microcirculatory) level, gas and nutrient exchange occurs, while macrocirculation facilitates these exchanges by ensuring that blood flows with appropriate pressure and velocity. A mismatch in this relationship, where the capillary perfusion does not correlate with the macrocirculatory parameters, is frequently observed in patients with shock or heart failure [3,4]. This discrepancy is often caused by capillary leak or hemodilution. To date, treatment has primarily focused on correcting macroscopically observed variables or values derived from them and resulting in pressure- or flow-dependent therapies.

While sublingual capillary perfusion measurements provide systemic insights, direct myocardial capillary perfusion assessment offers a direct and regional perspective. Unlike systemic capillary beds, myocardial perfusion is directly influenced by filling pressures, such as left ventricular end-diastolic pressure (LVEDP) [5]. Impaired myocardial capillary perfusion can lead to a cascade of cardiac dysfunction, including reduced oxygen delivery, inadequate nutrient exchange and making it vulnerable to ischemia or hibernation [1].

Current literature has examined intra- and postoperative sublingual (i.e., systemic) capillary perfusion following cardiac surgery [5]. Cardiopulmonary bypass (CPB), commonly used in many types of heart surgeries, inherently disrupts capillary perfusion due to its extracorporeal nature. The use of CPB alone triggers systemic inflammation, reperfusion injury and hemodilution, leading to the accumulation of metabolic waste products, formation of free oxygen radicals and perfusion alternations [7]. Additionally, the participants undergo an invasive cardiac procedure, accompanied by anesthesia and other contributing factors that negatively impact the capillary perfusion [8]. These alterations manifest in differences in microcirculatory parameters, including total vessel density (TVD), perfused vessel density (PVD), proportion of perfused vessels (PPV), microvascular flow index (MFI), and heterogeneity index (HI) [9].

Additionally, unloading the left ventricle (LV) unloading is posited to be critical for improving myocardial circulation. LV unloading is a promising concept that theoretically could improve capillary perfusion by reducing LVEDP and hence myocardial work. LV unloading could be particularly important for heart failure patients in acute cardiogenic shock. It may help promote myocardial circulation and prevent pulmonary edema. However, there is currently no robust scientific evidence to support these benefits and remains a subject of debate and philosophical discourse within the medical community [11-13].

To address this, the investigators aim to investigate whether capillary perfusion changes induced by CPB flow alterations, measured at sublingual and myocardial sites, provide consistent results. Additionally, the investigators will assess the effect of LV unloading on the capillary perfusion. The investigators will employ a handheld IDF-microcamera to perform real-time measurements of capillary perfusion. The investigators hypothesize that during hemodynamic alternations via CPB-flow sublingual and myocardial capillary perfusion measurements will show minimal differences and correlate with each other. This would supporting the validity of sublingual capillary perfusion measurements as a reliable, non-invasive proxy for the myocardial capillary perfusion status. Furthermore, the investigators anticipate an improvement in solely myocardial of both sublingual and myocardial capillary perfusion with LV unloading. These findings will significantly advance our understanding of the interaction between macro- and microcirculatory systems, providing a foundation for the use of sublingual measurements in both clinical and research settings. Ultimately, this could simplify monitoring techniques, enhance perioperative management, and help elucidate the mechanisms underlying persistent hemodynamic instability, guiding the development of more effective strategies to optimize postoperative outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older)
* Use of central cannulated CPB through median sternotomy
* Patients undergoing valve surgery or a supracoronary ascending aorta replacement
* Good LVEF and RVF
* LAVI < 50 ml/m2, and right atrial volume index (RAVI) < 45 ml/m2,

Exclusion Criteria:

* Patients with significant coronary artery disease (i.e., CAD-RADS ≥ 4, and/or stenosis of ≥ 70% as observed in coronary angiogram) or previous infarctions, including ST-elevated myocardial ischemia (STEMI) or non-ST-elevated myocardial ischemia (N-STEMI)
* Patients with echocardiographically observed regional wall motion abnormalities, hypokinesis, or akinesis in the coronary territories
* Patients undergoing left atrial appendage amputation (LAAA)
* Patients with AF
* High-risk patients, as defined by a EuroSCORE II ≥ 8%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients are selected from the surgical waiting list. Since we aim to include only elective adult patients with minimal comorbidities and a low or intermediate European System for Cardiac Operative Risk Evaluation (EuroSCORE) II (i.e., low or intermediate risk of in-hospital mortality), a significant number of patients are eligible. On our department, we perform approximately 20 cardiac surgeries per week, with valve surgeries representing a relatively large portion. The distribution of surgeries varies from week to week. However, a significant proportion of patients cannot be included due to the need for concomitant coronary revascularization or a history of such procedures
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
TVD (Total Vessel Density) | Intraoperatively
  The number of small blood vessels (< 20 μm) in a given area. (Vessel density in #/area)
PVD (Perfused Vessel Density) | Intraoperatively
  The number of small blood vessels that show perfusion, defined by a flow score of 2 or higher (moderate to normal flow). (Perfusion vessel density in #/area)
PVD (Perfused Vessel Density) | Intraoperatively
  The ratio of total vessel length to the length of perfused vessels. (Ratio)
MFI (Microvascular Flow Index) | Intraoperatively
  A semi-quantitative measure that evaluates flow in the capillary perfusion. (Flow score)
HI (Heterogenity Index) | Intraoperatively
  The degree of variation in capillary perfusion flow between different areas, calculated as the difference between the highest and lowest MFI, divided by the average MFI. (Variation index)

SECONDARY OUTCOMES:
Demographic information: Age | Preoperatively
  Reported in years.
Demographic Information: Gender | Preoperatively
  Categorized as male/female/other.
Demographic Information: Body Mass Index (BMI) | Preoperatively
  Calculated as weight (kg) divided by height squared (m²). Reported in kg/m²
Demographic Information: Medical History | Preoperatively
  Presence or absence of pre-existing conditions, such as hypertension, diabetes, prior heart surgeries; each condition reported as a separate categorical variable (yes/no).
Demographic Information: Comorbidities | Preoperateively
  Presence or absence of vascular disease other than coronary artery disease, kidney dysfunction, pulmonary disease; each as separate categorical variables.
Surgical Variables: Type of Underlying Pathology | Preoperatively
  Described separately for valve regurgitation, valve stenosis, aneurysm; categorical variable.
LV Unloading Variables: TVD (Total Vessel Density, # vessels per area) | Intraoperatively
  Capillary perfusion parameters measured separately, as they have different units and scales, consistent with primary objectives:
  Each perfusion parameter is reported separately for conditions with and without LV unloading.
LV Unloading Variables: PVD (Perfused Vessel Density, # vessels per area) | Intraoperatively
  Capillary perfusion parameters measured separately, as they have different units and scales, consistent with primary objectives:
  Each perfusion parameter is reported separately for conditions with and without LV unloading.
LV Unloading Variables: PPV (Proportion of Perfused Vessels, ratio) | Intraoperatively
  Capillary perfusion parameters measured separately, as they have different units and scales, consistent with primary objectives:
  Each perfusion parameter is reported separately for conditions with and without LV unloading.
LV Unloading Variables: MFI (Microvascular Flow Index, semi-quantitative score) | Intraoperatively
  Capillary perfusion parameters measured separately, as they have different units and scales, consistent with primary objectives:
  Each perfusion parameter is reported separately for conditions with and without LV unloading.
LV Unloading Variables: - HI (Heterogeneity Index, variation ratio) | Intraoperatively
  Capillary perfusion parameters measured separately, as they have different units and scales, consistent with primary objectives:
  Each perfusion parameter is reported separately for conditions with and without LV unloading.

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the outcome